CLINICAL TRIAL: NCT04715503
Title: PET-imaging of Unruptured Intracranial Aneurysm Inflammation
Acronym: PET-IA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Jaakko Rinne, Professor, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T225/2020
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Intracranial Aneurysm; Cerebral Aneurysm; Inflammation
Keywords: intracranial aneurysm; PET; inflammation; positron emission tomography; rupture risk
MeSH Terms: conditions — Intracranial Aneurysm; Inflammation | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18; 68Ga-DOTANOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET-IA (Experimental): 68Ga-DOTANOC 18F-FDG
  Interventions: Radiation: PET imaging, 18F-FDG; Radiation: PET imaging, 68Ga-DOTANOC

INTERVENTIONS:
Radiation: PET imaging, 18F-FDG — PET-MRI with 18F-FDG
Radiation: PET imaging, 68Ga-DOTANOC — PET-CT with 68Ga-DOTANOC

SUMMARY:
The main purpose of this study is to determine if PET-imaging can be used to evaluate inflammation level of intracranial aneurysms, thus helping to evaluate the rupture risk of intracranial aneurysm.

DETAILED DESCRIPTION:
Study subjects are patients who are diagnosed with an unruptured saccular intracranial aneurysm and planned for elective surgical treatment of intracranial aneurysms. Prior the planned surgery, all study subjects will undergo PET-imaging of the brain with 18F-FDG- and 68Ga-DOTANOC-tracers targeting glucose metabolism and somatostatin receptors in inflammatory cells. After PET-imaging, samples for histopathological examination from the intracranial aneurysm sac will be collected during the surgery from every study subject. Blood samples are collected prior to aneurysm operation from the routine pre-operative laboratory tests. Cerebrospinal fluid samples are collected during the surgical procedure from the surgical site. From blood samples we will evaluate expression of 20 different circulating microRNAs (miRNA) and the level of tumor necrosis factor-1, interleukin 1 beta, vascular endothelial growth factor, and evaluate correlations between miRNA expression and SUVmax in PET-imaging and miRNA and aneurysm histological findings.

Correlation between inflammatory findings in histological studies and PET-imaging will be evaluated (correlation of SUVmax to aneurysm histological findings).

ELIGIBILITY:
Inclusion Criteria:

* Fusiform intracranial aneurysms
* Following medications: Asetylsalisylic acid or non-steroidal anti-inflammatory drugs.
* Patients who have contraindication for magnetic resonance imaging (Pace Makers, foreign ferromagnetic bodies or implants)
* Patients who are allergic to contrast agents.
* Pregnancy
* Underage persons
* Patients on somatostatin analogue medication or with known neuroendocrine tumor

Exclusion Criteria:

* Patients who are diagnosed with unruptured intracranial aneurysm with MRI/MRA or DSA
* Patients who are planned to undergo surgical treatment (ligation) of the intracranial aneurysm
* Age ≥18 and <75 years.
* Saccular intracranial aneurysm with maximum diameter ≥ 3 mm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
PET-imaging of unruptured intracranial aneurysms | 1 month
  Uptake of 18F-FDG or 68Ga-DOTANOC in intracranial arterial aneurysms as compared to contra-lateral normal vessel as SUVmax or TBR.
  Correlation of uptake of 18F-FDG or 68Ga-DOTANOC (SUVmax or TBR) to aneurysm histological findings (CD45, CD3, CD5, CD20, CD138 and CD68, SSTR2, SSTR3 and SSTR5)

SECONDARY OUTCOMES:
Risk factors for intracranial aneurysm inflammation | 1 month
  Uptake of 18F-FDG or 68Ga-DOTANOC and histological findings correlation to aneurysm size and shape, smoking, hypertension, location of aneurysm.

CONTACTS AND LOCATIONS:
Overall Officials: Jaakko Rinne, MD, Prof., Principal Investigator — Turku University Hospital, Neurocenter, Department of Neurosurgery, Division of Clinical Neurosciences, University Of Turku; Antti Saraste, MD, Prof., Study Director — Turku University Hospital, Heart Centre, University of Turku
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Laukka D, Paturi J, Rahi M, Saraste A, Parkkola R, Kivelev J, Gardberg M, Kuhmonen J, Rinne J. PET imaging of unruptured intracranial aneurysm inflammation (PET-IA) study: a feasibility study protocol. BMJ Open. 2024 Feb 20;14(2):e076764. doi: 10.1136/bmjopen-2023-076764. PMID 38382960